CLINICAL TRIAL: NCT02849522
Title: ROPE Registry Project to Determine the Safety and Efficacy of Prostate Artery Embolisation (PAE) for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Enlargement (LUTS BPE).
Acronym: UKROPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cedar, United Kingdom (Other)
Collaborators: National Institute for Health and Care Excellence (NICE) (Unknown); British Society of Interventional Radiologists (BSIR) (Unknown); British Association of Urological Surgeons (BAUS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: UKROPE Register Study
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Lower Urinary Tract Symptoms Caused by Benign Prostatic Enlargement (LUTS BPE); Prostate Artery Embolisation (PAE); Transurethral Resection of the Prostate (TURP); Open Prostatectomy; Laser Enucleation or Ablation of the Prostate
Keywords: Lower Urinary Tract Symptoms caused by Benign Prostatic Enlargement (LUTS BPE); Prostate Artery Embolisation (PAE); Transurethral Resection of the Prostate (TURP); Open prostatectomy; Laser enucleation or ablation of the prostate (Green Light, KTP, HoLEP); IPSS Score; IIEF Score; Complications; Quality of Life
MeSH Terms: interventions — Transurethral Resection of Prostate; Laser Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PAE patients: Men who have undergone PAE and are in the UK ROPE Register
  Interventions: Procedure: Prostatic Artery Embolisation
- Comparator treatment patients: Men who have undergone TURP, Open Prostatectomy or laser ablation/enuclation of the prostate, and are on the UK ROPE Register.
  Interventions: Procedure: TURP; Procedure: Open prostatectomy; Procedure: Laser prostate surgery

INTERVENTIONS:
Procedure: Prostatic Artery Embolisation — The aim of PAE for LUTS (due to BPH) is to reduce the blood supply of the prostate gland, causing some of it to undergo necrosis with subsequent shrinkage.
  The procedure is usually performed with the patient under local anaesthetic and sedation. Using a percutaneous transfemoral approach, super-selective catheterisation of small prostatic arteries is carried out using microcatheters. Embolisation involves the introduction of microparticles to block these small prostatic arteries. Embolisation agents include polyvinyl alcohol (PVA), gelatine sponge and other synthetic biocompatible materials.
  NICE published Interventional Procedures Guidance (IPG453) in April 2013. The evidence at the time of assessment was deemed inadequate in quantity and quality. Therefore, the procedure was given a 'Research-only' recommendation.
  Groups: PAE patients
Procedure: TURP — Transurethral resection of the prostate. A cystoscope is passed up the urethra to the prostate, where the surrounding prostate tissue is excised. This is a common operation for benign prostatic hyperplasia (BPH), with around 15,000 procedures performed in the UK per year (NHS Choices). The conventional TURP method of tissue removal utilizes a wire loop with electrical current flowing in one direction (monopolar) through the resectoscope to cut the tissue. Bipolar TURP allows saline irrigation and eliminates the need for an ESU grounding pad thus preventing TUR syndrome and reducing other complications.
  Other Names: Transurethral resection of the prostate
  Groups: Comparator treatment patients
Procedure: Open prostatectomy — In an open prostatectomy the prostate is accessed through an incision that allows manual manipulation and open visualization through the incision. The most common types of open prostatectomy are retropubic prostatectomy (RP) or transvesical prostatectomy (TVP).
  Groups: Comparator treatment patients
Procedure: Laser prostate surgery — This surgical method (HoLEP or KTP/"Greenlight") utilizes laser energy to remove tissue. With laser prostate surgery a laser fibre inserted via an endoscope is used to transmit laser energy to enucleate (HoLEP) or vaporise (KTP) the tissue. The specific advantages of utilizing laser energy rather than a traditional electrosurgical TURP is a decrease in the relative blood loss, elimination of the risk of TUR syndrome, the ability to treat larger glands, as well as treating patients who are actively being treated with anti-coagulation therapy for unrelated diagnoses.
  Other Names: HoLEP; KTP; GreenLight; Laser ablation; Laser enucleation
  Groups: Comparator treatment patients

SUMMARY:
This is a study protocol for the UK ROPE Register for Lower Urinary Tract Symptoms (LUTS). This register enables us to collect data on the treatment of LUTS using prostate artery embolisation (PAE), and other surgical methods to answer the following questions posed by NICE in 2013:

* Is PAE a safe and effective treatment option for LUTS caused by prostate enlargement?
* How does PAE compare with conventional surgical treatments? This will primarily be a surgical procedure called TURP (see below).
* Which patients would most benefit from PAE over the other treatment options? This is a pilot study, and the final register will contain data from roughly 100 patients for PAE and 100 patients for the other surgical interventions, allowing us to answer NICE's research questions, update NICE guidance documentation, and do further research with more patients if necessary.

Our hypothesis is:

• PAE produces significant improvements in the IPSS score 12 months post-procedure

DETAILED DESCRIPTION:
This is a pilot study, intended to collect observational data on the PAE procedure as it is disseminated and performed around the UK, and on other comparator interventions. The aim is to give NICE enough information to potentially update their Interventional Procedures Guidance and may form the grounding for further research in the shape of a larger randomised clinical trial.

The ROPE Register project aims are to:

Primary:

• Assess the efficacy of PAE using the IPSS for LUTS BPE 12 months post-procedure.

Secondary:

* Compare PAE to TURP (using IPSS score) for LUTS BPE 12 months post-procedure. This will be a non-inferiority study for PAE versus TURP. A non-inferiority approach has been chosen because if PAE is no worse in terms of outcome for the patient, but is a more acceptable procedure to the patient (or has fewer complications, is less invasive, etc) than TURP, then PAE would be preferable.
* Use descriptive statistics for other outcome measures (IPSS, IPSS QoL, IIEF, prostate volume and urinary flow studies) for other comparator interventions (not TURP), 12 months post-procedure.
* Identify complications arising from PAE up to 12 months post-procedure.
* Elucidate which subgroup (s) of patients would benefit the most from PAE as a treatment option.

Our hypothesis is:

• PAE produces significant improvements in the IPSS score 12 months post-procedure

Additional subgroup analyses:

Other areas of interest from this research are covered in the subgroup analyses. The tables below detail the PAE patient subgroups that will be analysed. These subgroups will be cross-analysed with the measures in the Outcome measures table. This will enable trends to be noted in particular subgroups, which may inform future research.

Subgroups:

Age Baseline IPSS score Baseline Prostate Volume

Outcome measures:

IPSS Score IPSS Quality of Life Score IIEF score Prostate Volume Urinary flow study (Qmax, post-void residual volume, duration of micturition)

ELIGIBILITY:
Inclusion Criteria for this registry study:

* Men with LUTS who have consented for PAE, TURP, open prostatectomy or laser surgery at a participating site
* Able to read, write and understand English
* Capable of giving informed written consent

Exclusion Criteria for this registry study:

* Not able to read, write or understand English
* Not able/willing to provide informed written cons

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It should be noted that the dissemination of the PAE procedure in the UK is separate to this registry study. Therefore, the inclusion criteria for this registry study are all patients who have had PAE or one of the comparator interventions (TURP, open prostatectomy or laser surgery) in one of the participating hospitals. and outline of the inclusion/exclusion guidelines for participating hospitals is shown below:
  Inclusions for patient selection at participating hospital:
  Age 50-75 Moderate to severe LUTS Prostate volume ≥ 40 ml Maximum urinary flow rate < 12ml/s Unsuccessful drug therapy for ≥ 6 months
  Exclusions for patient selection at participating hospital:
  Atherosclerosis of the prostatic arteries Bladder diverticula or stone Urethral stenosis Neurogenic bladder eGFR ≤ 45ml min-1m-2 Malignancy (on biopsy)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
IPSS score change in PAE patients from baseline measurement | 12 months
  Assess the efficacy of PAE using the IPSS for LUTS BPE 12 months post-procedure.

SECONDARY OUTCOMES:
PAE non-inferiority to TURP 12 months post-procedure, using IPSS | 12 Months
  Compare PAE to TURP (using IPSS score) for LUTS BPE 12 months post-procedure. This will be a non-inferiority study for PAE versus TURP. A non-inferiority approach has been chosen because if PAE is no worse in terms of outcome for the patient, but is a more acceptable procedure to the patient (or has fewer complications, is less invasive, etc) than TURP, then PAE would be preferable.

OTHER OUTCOMES:
Identify complications arising from PAE up to 12 months post-procedure | 12 months
  Identify complications arising from PAE up to 12 months post-procedure
Subgroup analyses | 12 months
  Other areas of interest from this research are covered in the subgroup analyses, such as age or initial prostate volume. These subgroups will be cross-analysed with the various standard urological outcome measures such as Qmax and prostatic volume at 12 months post procedure. This will enable trends to be noted in particular subgroups, which may inform future research.
Descriptive statistics for other outcome measures | 12 months
  Use descriptive statistics for other urological outcome measures e.g. IPSS for other comparator interventions (not TURP), 12 months post-procedure.